CLINICAL TRIAL: NCT02800239
Title: Evaluation of Protein Requirements in Active Adolescent Females
Brief Title: Protein Requirements for Active Adolescent Females
Acronym: IAAO-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAAO-AF
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Increased Metabolic Requirement; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active, adolescent females (Experimental): Subjects will receive different levels of amino acid intakes, varying from 0.2-2.67 g/kg/d
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Amino acid intakes will be varied at 0.2-2.67 g/kg/d

SUMMARY:
Protein requirements in active individuals have been suggested to be greater than the current recommended dietary allowance (RDA).

Nutritional requirements for dietary amino acids in adolescents have traditionally been determined utilizing the nitrogen balance technique, which is prone to underestimating protein requirements. As a result, there is a need to re-evaluate recommendations in order to characterize how dietary amino acid needs may be modulated by physical activity.

Recent studies using the minimally invasive indicator amino acid oxidation (IAAO) technique have suggested that protein requirements in young men are at least 50% higher than the RDA based on nitrogen balance data.

The purpose of this study is to measure the protein requirement in adolescent, females using the IAAO technique in the presence of a variable intensity exercise stimulus.

ELIGIBILITY:
Inclusion Criteria (Adolescents):

* Healthy, active adolescent who regularly participates in moderate to vigorous physical activity 5 times a week for a minimum of 1 hour.
* Being -0.5 to +1.0 years from peak height velocity, determined by the ratio of standing to sitting height, with the maximal age for adolescents being 16 years.

Obtaining a minimum level of 5.8 on the Beep Test

Exclusion Criteria (All Subjects):

* Inability to meet health and physical activity guidelines according to the Physical Activity Readiness Questionnaire (PAR-Q+) and Physical Activity Questionnaire,
* An inability to adhere to any of the protocol guidelines (i.e. caffeine consumption)
* A biological age falling outside of the aforementioned ranges

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
13CO2 ([13]Carbon Dioxide) Excretion (µmol/kg/h) | 4 hours/ study day

SECONDARY OUTCOMES:
[13C]Phenylalanine Oxidation (µmol/kg/h) | 4 hours/ study day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No